CLINICAL TRIAL: NCT07022002
Title: A Phase II Study to Evaluate the Safety and Efficacy of SSGJ-705 Monotherapy and Combination Therapy in Patients With Advanced HER2-Expressing Solid Tumors
Brief Title: SSGJ-705 Monotherapy and Combination Therapy in Advanced HER2-Expressing Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-705-201
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced, Recurrent or Metastatic Malignancies
Keywords: advanced malignancies
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): advanced gastric cancer and breast cancer that have failed standard treatment
  Interventions: Drug: SSGJ-705
- Part 2 (Experimental): previously untreated advanced gastric cancer and lung cancer
  Interventions: Drug: PD-1/L1 inhibitor combined with chemotherapy; Drug: SSGJ-705 combined with chemotherapy

INTERVENTIONS:
Drug: SSGJ-705 — anti-PD-1 (programmed cell death protein 1) and anti-HER2 (Human Epidermal GrowthFactor Receptor 2)bispecifc antibody
  Arms: Part 1
Drug: PD-1/L1 inhibitor combined with chemotherapy — Immune checkpoint inhibitors
  Arms: Part 2
Drug: SSGJ-705 combined with chemotherapy — anti-PD-1 and anti-HER2 bispecifc antibody
  Arms: Part 2

SUMMARY:
This study was an open-label phase Ⅱ study to evaluate the safety and efficacy of SSGJ-705 Monotherapy and Combination Therapy in patients with advanced HER2-Expressing Solid Tumors.

DETAILED DESCRIPTION:
This study includes 2 Parts: Part 1 (705 monotherapy for advanced gastric cancer and breast cancer that have failed standard treatment), and Part 2 (705 in combination with chemotherapy for previously untreated advanced gastric cancer and lung cancer).

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females over age 18.
* Histologically and/or cytologically documented local advanced or metastatic non-Small Cell Lung Cancer（NSCLC），Breast Cancer（BC）or Gastric/Gastroesophageal Junction Cancer （G/GEJC).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival >3 months.
* Signed informed consent form.

Exclusion Criteria:

* Any remaining adverse events (AEs) > grade 1 from prior anti-tumor treatment as per Common Terminology Criteria for Adverse Events（CTCAE） v5. 0, with exception of hair loss, fatigue, and grade 2 peripheral neurotoxicity.
* Pregnant or nursing women or women/men who are ready to give birth.
* symptomatic central nervous system metastasis.
* Allergy to other antibody drugs or any excipients in the study drugs.
* Inadequate organ or bone marrow function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
  The primary efficacy end point
Incidence of Treatment-Emergent Adverse Events | 12 months
  The primary safety end point
Severity of Treatment-Emergent Adverse Events | 12 months
  The primary safety end point

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | 24 months
  The secondary efficacy end point

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No